CLINICAL TRIAL: NCT03713983
Title: Characteristics of and Treatment Outcomes Among Patients With Prescription Narcotic Drug Use Disorder: a Naturalistic Cohort Study
Brief Title: Treatment Outcomes Among Patients With Prescription Narcotic Drug Use Disorder
Acronym: TAPE
Status: Active, not recruiting | Type: Observational
Sponsor: Johan Franck (Other)
Collaborators: Public Health Agency of Sweden (Other Government)
Responsible Party: Sponsor-Investigator, Johan Franck, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: TAPE 2018
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Drug Use Disorders
Keywords: behavior, addictive; addiction medicine; substance-related disorders; abuse, narcotic; addiction, narcotic; analgesics, narcotic; opioid-related disorders; benzodiazepines; prescription drugs
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive; Narcotic-Related Disorders; Opioid-Related Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | US Export: No

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
This study follows up patients who receive standard treatment for prescription narcotic drug use disorder, including opioids, benzodiazepines, and benzodiazepine-like drugs (z-drugs), at a specialized addiction service. The overall goal is to evaluate the proportion of patients who reduce or cease using prescription narcotics and the factors associated with treatment outcomes. No new treatments will be tested. Instead, the results will be used as the basis for a future randomized controlled trial to optimize treatment for narcotic drug use disorder.

DETAILED DESCRIPTION:
Background: The study covers prescription narcotics and focuses on opioids and benzodiazepines (and related compounds). The use of opioids and benzodiazepines is relatively safe in the short term. However, long-term use for anxiety and chronic non cancer pain has limited scientific support. Moreover, use of opioids and benzodiazepines has been associated with a variety of adverse effects and both opioids and benzodiazepines are highly addictive.

Clinical guidelines advise that narcotic analgesics and sedatives should not be used as first-choice treatments for pain, anxiety, or insomnia. Instead, guidelines recommend psychotherapy, physiotherapy, and non-narcotic pharmacological drugs (such as non-steroidal anti-inflammatory drugs and antidepressants), alternatives that are less addictive and more beneficial over time. Despite such recommendations, benzodiazepines and opioids are commonly prescribed and used over the long term.

For patients who seek treatment for narcotic drug use disorder, tapering by gradual dose reduction is an important component but its effect is not well studied.

Aims: This study aims to investigate the clinical trajectory and treatment outcome among patients with narcotic drug use disorder at specialized addiction treatment services.

Specific aims:

1) The outcome of tapering of narcotic drugs at 6, 12, and 24 months follow-up 2) How the treatments provided (e.g., tapering; tapering plus psychological treatment) are associated with patient outcomes 3) How psychiatric symptoms and comorbidity are associated with patient outcomes 4) Predictors of narcotic drug abstinence and retention in treatment 5) The validity of psychiatric diagnoses in relation to drug use (i.e., whether the diagnosis changes significantly following drug detoxification)

Methods: This is a naturalistic, prospective study of outcomes following treatment at a specialized service for prescription narcotic drug use disorder. Standardized screening and assessment tools will be used to investigate patients at baseline, evaluate the treatment patients receive over a 24-month period, and evaluate patient outcomes.

All patients starting a new treatment period at the center will be invited to participate at the first visit to the clinic or as soon as possible thereafter. Written informed consent will be obtained. The study will conform to Good Clinical Practice (ICH-GCP) and the principles outlined in the Declaration of Helsinki.

Measurements in the study include: urine drug screening, blood chemistry including screening for alcohol biomarkers, Drug Use Disorders Identification Test, Alcohol Use Disorders Identification Test, Patient Health Questionnaire, EuroQol -5D, Clinical Global Impressions Scale, Adult ADHD Self-Rating Scale - Screening, The Mini International Neuropsychiatric Interview, Version 7, the Life Events Checklist, the Insomnia Severity Index, the Benzodiazepine Withdrawal Symptom Questionnaire, the Subjective Opioid Withdrawal Scale, Generalized Anxiety Disorder - 7, Numeric Rating Scale for Pain, PROMIS Pain Interference - Short Form 4a, patient satisfaction, Substance use questionnaire, and Structural Clinical Interview for DSM-IV Axis II Personality Disorders Screening.

Information regarding treatment at the unit (e.g. number and type of visits, somatic or psychiatric diagnoses) will be collected from medical records using the ICD codes. Diagnostic assessment will be performed according to both ICD-10 and DSM-5.

The protocol allows for a 10-year follow-up using national registries.

Study procedures and data collection will be regularly monitored by an external quality assurance organization.

Analyses will be conducted using statistical software; p values < 0.05 will be considered significant. Prescription drug use, retention in treatment and the percentage of participants with negative urine samples and self-reported abstinence will be calculated at follow-ups. Regression analyses will be computed to assess factors associated with the outcome of tapering.

To find a 95 % confidence interval around the point estimate (drug abstinence) with a margin of error not exceeding +/- 5 percentage points, where the assumed proportion is 0.3, at least 322 patients must be included. Alternatively, to find a 95 % confidence interval with a margin of error not exceeding +/- 10 percentage points, at least 81 patients must be included. A minimum of 81 patients will be included in the study. The study will include an analysis of dropout.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking treatment for prescription narcotic drug use disorder (ICD-10: F111, F112, F131, and F132)
* ≥ 18 years
* Willing to participate and who have provided written informed consent.

Exclusion Criteria:

* Inability to understand spoken and written study information.
* Having started tapering prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients starting a new treatment period for prescription narcotic drug use disorder
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in prescription narcotic drug use | 6-, 12- and 24-month follow-up or at last visit; 10-year follow-up.
  Change in dosage of prescription narcotic drugs

SECONDARY OUTCOMES:
Prescription narcotic drug abstinence | 6-, 12- and 24-month follow-up or at last visit
  Measured by drug testing and self-reported substance use
Retention in treatment | 6-, 12- and 24-month follow-up or at last visit
  Data collected from scheduled visit

OTHER OUTCOMES:
Diagnoses of substance use disorder(s) | 6-, 12-, and 24-month follow-up
  Number of participants with diagnoses of substance use disorder according to ICD-10
Self-reported substance use | 6-, 12-, and 24 month follow-up
  self-reported data using standard question in ASI
Psychiatric comorbidity | 6-, 12-, and 24-month follow-up
  Number of participants with psychiatric diagnoses according to ICD-10
Personality traits | 6-, 12-, and 24-month follow-ups
  SCID-2 Structured Clinical Interview for DSM-IV-Axis 2 Disorders, screening
Insomnia | 6-, 12-, and 24-month follow-up
  Insomnia Severity Index (ISI)
Pain Scale | 6-, 12-, and 24-month follow-up
  The PROMIS pain interference - Short form 4a (PROMIS-PI SF 4a), is a four-item questionnaire measuring the extent pain interferes with functioning in daily life. Items are rated on a five-point scale ranging from "not at all" to "very much". Summed scores range from 4-20, higher scores indicating greater pain interference. The scale is recommended by the National Institute of Drug Abuse (NIDA).
Quality of life, including self-rated health | 6-, 12-, and 24-month follow-up
  Measured by EuroQol 5D (EQ-5D), a two-part health index. Part one covers self-rated problems in five domains: mobility, self-care, everyday activities, pain/discomfort, and anxiety/depression. Each domain is rated on a five-level scale that indicates no problems to extreme problems. Part two consist of a visual analog scale (EQ-5D VAS); respondents assess their subjective health status on a 0 to 100 scale, where 0 is "the worst health you can image" and 100 "the best health you can imagine."
Somatic health | 6-, 12-, and 24-month follow-up
  Number of participants with somatic diagnoses according to ICD-10
Withdrawal symptoms Opioids | 6-, 12-, and 24-month follow-up
  Measured by the Subjective Opiate Withdrawal Scale (SOWS). The scale measures 16 common symptoms of opiate withdrawal. Symptoms are rated on a scale between 0 and 4, from "not at all" to "extremely." Higher scores indicating more withdrawal symptoms.
Substitution treatment with opioids | 6-, 12-, and 24-month follow-up
  Prescription registry data
Withdrawal symptoms Benzodiazepines | 6-, 12-, and 24-month follow-up
  The Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ)
Self-reported patient satisfaction with treatment | 6-, 12-, and 24-month follow-up
  Self-report data using standard question in the National Patient Survey (Sweden). Items measures patients' experience and satisfaction with care. Items are rated on a scale between 1 ("Not at all") and 5 ("Totally agree"), with the possibility to answer "Not applicable".

CONTACTS AND LOCATIONS:
Overall Officials: Johan Franck, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm Centre for Dependency Disorders (www.beroendecentrum.se), Stockholm, Sweden

REFERENCES:
- [Derived] Burmester S, Kruger C, Hallgren J, Westman J, Franck J. A prospective cohort of treatment-seeking patients with problematic use of prescription narcotic drugs: study protocol and baseline characteristics. BMC Psychiatry. 2024 Dec 20;24(1):937. doi: 10.1186/s12888-024-06368-w. PMID 39707239